CLINICAL TRIAL: NCT01967862
Title: F18 NaF PET/CT and Whole Body and Axial MRI for the Detection of Metastases in Patients With Biochemical Recurrence of Prostate Cancer
Brief Title: Fluorine F 18 Sodium Fluoride PET/CT and Whole Body and Axial MRI in Finding Metastases in Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13365; NCI-2013-01924 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13365 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2018-09

CONDITIONS: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (CT, bone scan, WB/axial MRI, F18 NaF PET/CT) (Experimental): Patients first undergo CT scan and bone scan. Patients with negative results from the CT and bone scans then undergo WB MRI scan using diffusion-weighted MRI, axial MRI scan using 3-Tesla MRI, and fluorine F 18 sodium fluoride PET/CT scan.
  Interventions: Procedure: computed tomography; Procedure: bone scan; Procedure: 3-Tesla magnetic resonance imaging; Procedure: diffusion-weighted magnetic resonance imaging; Radiation: fluorine F 18 sodium fluoride; Procedure: positron emission tomography; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: computed tomography — Undergo CT
  Other Names: tomography, computed
Procedure: bone scan — Undergo bone scan
Procedure: 3-Tesla magnetic resonance imaging — Undergo axial MRI
  Other Names: 3-Tesla MRI; 3T MRI
Procedure: diffusion-weighted magnetic resonance imaging — Undergo WB MRI
  Other Names: diffusion-weighted MRI
Radiation: fluorine F 18 sodium fluoride — Undergo fluorine F 18 sodium fluoride PET/CT
  Other Names: 18 F-NaF; F-18 NaF
Procedure: computed tomography — Undergo fluorine F 18 sodium fluoride PET/CT
  Other Names: tomography, computed
Procedure: positron emission tomography — Undergo fluorine F 18 sodium fluoride PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well fluorine F 18 sodium fluoride positron emission tomography (PET)/computed tomography (CT) and whole body and axial magnetic resonance imaging (MRI) work in finding metastases in patients with recurrent prostate cancer. New imaging techniques, such as fluorine F 18 sodium fluoride PET/CT and whole body and axial MRI, may be more effective than standard CT and bone scan in finding metastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients with biochemically-recurrent prostate cancer (PC) in whom imaging with whole body (WB)/axial MRI and F-18 NaF (fluorine F 18 sodium fluoride) PET/CT results in detection of metastatic disease not visualized on CT scan and bone scan.

SECONDARY OBJECTIVES:

I. To estimate the percent of eligible patients with negative, indeterminate and positive CT scan/bone scan and targeted X-rays if done.

II. To determine the proportion of patients with biochemically-recurrent PC in whom recurrence in the prostate bed can be visualized using MRI in the absence of detection using CT scan.

III. To correlate the presence of metastatic disease detected using WB/axial MRI and/or F-18 NaF PET/CT with the predicted 6-year probability of progression-free survival based on the Memorial Sloan Kettering Cancer Center salvage radiation therapy (RT) PC nomogram, and with prostate-specific antigen (PSA) level at baseline.

IV. To compare the role of axial MRI of the spine to WB/axial MRI with respect to their ability to identify sites of disease. Similarly, to evaluate the relative contribution of F-18 NaF PET and WB/axial MRI.

OUTLINE:

Patients first undergo CT scan and bone scan. Patients with negative results from the CT and bone scans then undergo WB MRI scan using diffusion-weighted MRI, axial MRI scan using 3-Tesla MRI, and fluorine F 18 sodium fluoride PET/CT scan.

After completion of study, patients are followed up at 4-6 months and periodically until week 52.

ELIGIBILITY:
Inclusion Criteria:

* History of prior radical prostatectomy for prostate cancer
* Two PSA values >= 0.2 ng/mL at least 4 weeks after prostatectomy
* Patients who have started radiographic evaluation and underwent CT scan and/or bone scan prior to registration to the study will be able to participate under a late registration provision, provided that the more modern scans (WB/axial MRI and F-18 NaF PET/CT) can be completed within 8 weeks after CT scan and bone scan

Exclusion Criteria:

* Patients with known metastatic disease
* PSA recurrence not verified by elevated PSA as discussed in the eligibility section
* Patients who initiated androgen deprivation therapy or other systemic therapy (chemotherapy, immunotherapy, targeted therapy) for PSA recurrence; nutritional supplements used for treatment of PSA recurrence will be allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-12; Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cy Stein, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (CT, Bone Scan, WB/Axial MRI, F18 NaF PET/CT)
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (CT, Bone Scan, WB/Axial MRI, F18 NaF PET/CT)
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 10
  Caucasian | 34
  African American | 4
  Asian | 6
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Patients With Positive CT Scan/Bone Scan, MRI and PET Scan.
Description: Count of eligible patients with positive CT chest, abdomen, pelvis scan, positive WB/axial MRI, positive F-18 NaF PET/CT and positive Bone scan for detection of metastatic disease.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (CT, Bone Scan, WB/Axial MRI, F18 NaF PET/CT)
Number analyzed (Participants) | 54
Participants
  Positive CT Scan | 0
  Positive Bone Scan | 0
  Positive MRI | 12
  Positive PET | 17

ADVERSE EVENTS:
Time Frame: Adverse Event occurred over a period of 1 year and 10 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Diagnostic (CT, Bone Scan, WB/Axial MRI, F18 NaF PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 4/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (CT, Bone Scan, WB/Axial MRI, F18 NaF PET/CT) (N=54)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatic lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT01967862/Prot_SAP_000.pdf